CLINICAL TRIAL: NCT03026231
Title: A Prospective, Randomized Placebo Controlled Pilot Study to Characterize the Intestinal Microbiome and to Evaluate the Safety and Fecal Microbiome Changes Following Weekly Administration of Lyophilized PRIM-DJ2727 Given Orally in Subjects With Parkinson's Disease
Brief Title: Characterization of Fecal Microbiome Changes After Administration of PRIM-DJ2727 in Parkinson's Disease Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study will be started under a new modified protocol
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Kelsey Research Foundation (Other)
Responsible Party: Principal Investigator, Herbert DuPont, Professor of Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UT-SPH/KRF FMT-2016-PD-01
Record Dates: First submitted 2017-01-11; First posted 2017-01-20 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
Keywords: Fecal microbiota transplantation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRIM-DJ2727 (Active Comparator): Subjects with PD will be randomly assigned to receive PRIM-DJ2727 in orally administered enteric-coated capsules
  Interventions: Biological: PRIM-DJ2727
- Placebo (Placebo Comparator): Thirty eligible subjects with PD will be randomly assigned to receive placebo capsules
  Interventions: Drug: Placebo (for PRIM-DJ2727)

INTERVENTIONS:
Biological: PRIM-DJ2727 — Thirty eligible subjects with PD will be randomly assigned to receive either PRIM-DJ2727 in orally administered enteric-coated capsules or placebo capsules
  Arms: PRIM-DJ2727
Drug: Placebo (for PRIM-DJ2727) — Thirty eligible subjects with PD will be randomly assigned to receive placebo capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the intestinal flora in subjects with Parkinson's Disease (PD) and to determine safety and trends in improvements in diversity of colonic microbiome following fecal microbiota transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis PD with a Hoehn and Yahr stage of < 3 in the "Off medicine" state
* Sexually active male and female subjects of child-bearing potential must agree to use an effective method of birth control during the treatment and follow-up period
* Female subjects of child-bearing potential must have a negative pregnancy test in the 72 hours before the procedure
* Subject willing to sign an informed consent form
* Subject deemed likely to survive for ≥ 1 year after enrolment
* Subject's attending physician will refer and provide non-transplant care for the subject
* Subjects must demonstrate adherence to and the ability to maintain a Parkinson's therapy medical regimen that is stable for 90 days before enrolment and participation in the study.

Exclusion Criteria:

* Greater than 20 grams of ethanol intake daily
* Unstable Parkinson's disease
* Other immune disorder or clinical immunosuppression
* Probiotic used during study period
* Severe underlying disease such that the subject is not expected to survive for one or more years or unstable medical condition requiring frequent change in treatments
* Current or recent within one month receipt of an antibiotic with expected activity against enteric bacteria
* Prior Deep Brain Stimulation, or surgical intervention for PD , intravenous glutathione therapy or stem cell therapy
* HIV or Hepatitis B / C positive

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Microbiome Diversity in Fecal Samples s Indicated by the Shannon Diversity Index | 3 years
Microbiome Diversity in Fecal Samples s Indicated by the Shannon Diversity Index | 6 months
Microbiome Diversity in Fecal Samples s Indicated by the Shannon Diversity Index | 12 months
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | 3 years
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | 6 months
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | 12 months
Most abundant Phylum in Fecal Sample | 3 years
Most abundant Phylum in Fecal Sample | 6 months
Most abundant Phylum in Fecal Sample | 12 months

SECONDARY OUTCOMES:
Improvements in flora diversity by oral administration of a fecal suspension from healthy donors comparing data with untreated controls | 3 years
Number of bowel movements per day | 3 years
Number of bowel movements per day | 6 months
Number of bowel movements per day | 12 months
Neurologic functioning as indicated by score on the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 3 years
  The (MDS-UPDRS) measures mentation, behaviour, mood, activities of daily living and motor manifestations and the Montreal Cognitive Assessment (MoCA) for memory assessment.
Neurologic functioning as indicated by score on the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 1 day
  The (MDS-UPDRS) measures mentation, behaviour, mood, activities of daily living and motor manifestations and the Montreal Cognitive Assessment (MoCA) for memory assessment.
Neurologic functioning as indicated by score on the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 6 months
  The (MDS-UPDRS) measures mentation, behaviour, mood, activities of daily living and motor manifestations and the Montreal Cognitive Assessment (MoCA) for memory assessment.
Neurologic functioning as indicated by score on the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 12 months
  The (MDS-UPDRS) measures mentation, behaviour, mood, activities of daily living and motor manifestations and the Montreal Cognitive Assessment (MoCA) for memory assessment.
Number of participants with a change in required anti-PD symptomatic or levodopa therapy | 12 months
Subject assessment of global improvement in PD and quality of life as indicated by score the self-survey Parkinson's Disease Questionnaire 39 (PDQ-39) | 3 years
Subject assessment of global improvement in PD and quality of life as indicated by score the self-survey Parkinson's Disease Questionnaire 39 (PDQ-39) | day 1 of treatment
Subject assessment of global improvement in PD and quality of life as indicated by score the self-survey Parkinson's Disease Questionnaire 39 (PDQ-39) | 6 months
Subject assessment of global improvement in PD and quality of life as indicated by score the self-survey Parkinson's Disease Questionnaire 39 (PDQ-39) | 12 months
Memory as assessed by score on the Montreal Cognitive Assessment (MoCA) | 3 years
Memory as assessed by score on the Montreal Cognitive Assessment (MoCA) | day 1 of treatment
Memory as assessed by score on the Montreal Cognitive Assessment (MoCA) | 6 months
Memory as assessed by score on the Montreal Cognitive Assessment (MoCA) | 12 months
Number of participants with worsening of PD symptoms or other potential flora-mediated disorders as indicated by patient diares | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L DuPont, MD, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Background] Borody TJ, Paramsothy S, Agrawal G. Fecal microbiota transplantation: indications, methods, evidence, and future directions. Curr Gastroenterol Rep. 2013 Aug;15(8):337. doi: 10.1007/s11894-013-0337-1. PMID 23852569
- [Background] Fasano A, Bove F, Gabrielli M, Petracca M, Zocco MA, Ragazzoni E, Barbaro F, Piano C, Fortuna S, Tortora A, Di Giacopo R, Campanale M, Gigante G, Lauritano EC, Navarra P, Marconi S, Gasbarrini A, Bentivoglio AR. The role of small intestinal bacterial overgrowth in Parkinson's disease. Mov Disord. 2013 Aug;28(9):1241-9. doi: 10.1002/mds.25522. Epub 2013 May 27. PMID 23712625
- [Background] Nakane S, Yoshioka M, Oda N, Tani T, Chida K, Suzuki M, Funakawa I, Inukai A, Hasegawa K, Kuroda K, Mizoguchi K, Shioya K, Sonoda Y, Matsuo H. The characteristics of camptocormia in patients with Parkinson's disease: A large cross-sectional multicenter study in Japan. J Neurol Sci. 2015 Nov 15;358(1-2):299-303. doi: 10.1016/j.jns.2015.09.015. Epub 2015 Sep 8. PMID 26428310